CLINICAL TRIAL: NCT06906302
Title: Recovering From IPV Through Strengths and Empowerment (RISE) Versus Advocacy-based Enhanced Care as Usual for Patients Experiencing IPV
Brief Title: RISE Versus Advocacy-based Enhanced Care as Usual for Patients Experiencing IPV
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); VA Philadelphia Healthcare System (Unknown); VA Minnesota Healthcare System (Unknown); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-45215; BPS-2023C2-33320 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2025-04-01; First posted 2025-04-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Intimate Partner Violence (IPV)
Keywords: RISE; Enhanced Care as Usual (ECAU); Healthcare patients; Self-efficacy; Depression; Post-Traumatic Stress Disorders (PTSD)
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RISE (Recovering from Intimate Partner Violence through Strengths and Empowerment) (Experimental): Participants randomized to the RISE arm will have 1 or more RISE sessions.
  Interventions: Behavioral: RISE
- Advocacy-based ECAU (Enhanced Care as Usual) (Active Comparator): Participants randomized to this arm will have a single Advocacy-based ECAU session
  Interventions: Behavioral: Advocacy-based ECAU

INTERVENTIONS:
Behavioral: RISE — RISE is personalized, trauma-informed, empowerment-oriented and variable-length, consisting of an initial 60-minute session and up to 7 additional 45-minute sessions (1-8 sessions total).
  Arms: RISE (Recovering from Intimate Partner Violence through Strengths and Empowerment)
Behavioral: Advocacy-based ECAU — Advocacy-based ECAU is a single 60-minute trauma-informed counseling intervention that includes supportive education, validating and empathetic statements, safety planning, resource provision and referrals.
  Arms: Advocacy-based ECAU (Enhanced Care as Usual)

SUMMARY:
This study aims to improve treatment for Veterans Health Administration (VHA) patients who experience intimate partner violence (IPV). This study will evaluate two brief counseling interventions for VHA patients who have experienced IPV in the past 12 months: Recovering from IPV through Strength and Empowerment (RISE) and advocacy-based Enhanced Care as Usual (ECAU). The RISE intervention includes up to 8 sessions and includes specific topic areas (e.g., social support, health effects, resources). The other intervention, ECAU, includes a single session that includes supportive education about IPV and health effects, discussion of ways to increase safety, and information about resources. This study will test which approach is better for improving self-efficacy and other aspects of health.

Participants will answer surveys about their self-efficacy and other health and safety indicators (e.g., mental health symptoms) right before receiving treatment, approximately 12 weeks later, and then every three months after that for one year. Participation in this research will last about 15 months.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving care at an enrolled site/affiliated Community-Based Outpatient Clinic (CBOC)
* report experience of past-year physical, psychological, and/or sexual IPV on an established screening tool used to detect IPV in VHA, and
* be able to provide informed consent including permission to have intervention sessions recorded

Exclusion Criteria:

* severe cognitive impairment,
* suicide or homicide intent with a specific plan
* untreated or unstable symptoms of mania or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy | Baseline, 3 months, 6 months. 9 months, 12 months, 15 months
  Self-efficacy will be assessed with the General Self-Efficacy Scale (GSES), a 10-item instrument with possible responses for each item from 1 to 4 where 1= Not at all true, 2= Hardly true, 3= Moderately true, and 4=Exactly true.Scores can range from 10 to 40 and higher scores indicate more self efficacy.

SECONDARY OUTCOMES:
Depressive symptoms | Baseline, 3 months, 6 months. 9 months, 12 months, 15 months
  Depressive symptoms will be assessed with the Center for Epidemiologic Studies Depression Scale (CESD), a 20-item instrument with possible responses for each item from 0 to 3 where 0= Rarely or none of the time (less than 1 day), 1= Some or a little of the time (1-2 days), 2= Occasionally or a moderate amount of the time (3-4 days), and 3= Most or all of the time (5-7 days). Possible range of scores is 0 to 60, with the higher scores indicating more depressive symptoms.
Post traumatic stress disorder (PTSD) symptoms | Baseline, 3 months, 6 months. 9 months, 12 months, 15 months
  PTSD symptoms will be assessed with the PTSD Checklist -DSM-5, a 20-item self-report measure of the DSM-5 symptoms of PTSD. A 5-point Likert scale is used for each item from 0 = "Not at all" to 4 = "Extremely". Total possible scores can range from 0 to 80 with higher scores indicating more PTSD symptoms.
Alcohol use | Baseline, 3 months, 6 months. 9 months, 12 months, 15 months
  Alcohol use will be assessed with the Alcohol Use Disorders Identification Test-10 (AUDIT-10), a 10-item instrument with possible responses for each item from 0 to 4 for questions 1-8 and possible responses of 0, 2, and 4 for questions 9 and 10. Total possible scores can range from 0 to 40 with higher scores indicating greater alcohol use.
Hopelessness | Baseline, 3 months, 6 months. 9 months, 12 months, 15 months
  Hopelessness will be assessed by the 20-item Beck Hopelessness Scale (BHS). The BHS is scored by adding up the responses to 20 true-false questions. The possible score range is 0-20, with higher scores indicating greater hopelessness.
Self-reported quality of life | Baseline, 3 months, 6 months. 9 months, 12 months, 15 months
  Quality of life will be assessed by World Health Organization - Quality of Life, Brief WHOQOL-BREF instrument, a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale with higher scores indicating a better quality of life.
Valued living | Baseline, 3 months, 6 months. 9 months, 12 months, 15 months
  Valued living will be assessed with the Valued Living Questionnaire (VLQ) focusing on 10 valued domains of living which include (1) family, (2) marriage/couples, intimate relations, (3) parenting, (4) friendship, (5) work, (6) education, (7) recreation, (8) spirituality, (9) citizenship, and (10) physical self-care. Each domain is rated on a scale of 1-10, based on the level of importance to the respondent and the extent to which they have lived consistent with their values in the past week. A total score is calculated by multiplying the importance and consistency ratings for each domain, and then averaging those scores. Total scores range from 10 to 100 with higher scores indicating greater alignment with one's values.
IPV | Baseline, 3 months, 6 months. 9 months, 12 months, 15 months
  Experiences of IPV from past or a current intimate partner will be measured using subscales of the Revised Conflict Tactics Scale (CTS-2). The physical aggression (12 items), psychological aggression (8 items), and sexual coercion (7 items) subscales include 27 items regarding the frequency of different IPV experiences (0=this has never happened, 1=1 time, 2=2 times, 3=3-5 times, 4=6-10 times, 5=11-20 times, and 6=20+ times). Items are summed for a total frequency score. Additionally, the number of different IPV behaviors experienced can be tallied to reflect a indicate the number of different IPV behaviors experienced. Higher scores reflect greater levels of IPV experience.
Measure of Victim Empowerment Related to Safety | Baseline, 3 months, 6 months. 9 months, 12 months, 15 months
  Safety-related Empowerment will be measured with the Measure of Victim Empowerment Related to Safety (MOVERS), a 13- item measure that consists of three subscales: internal resources (6 items), expectations of support (4 items), and trade-offs (3 items), with response options on a scale from 1-5, with 1 being "never true" and 5 being "always true" for each internal resource and expectation of support subscale question. Responses options for the trade-off subscale are reverse scored with 1 = Always true and 5= Never true. Total possible scores can range from 13 to 65, with higher scores indicating higher levels of empowerment.
Health care and social service use | Baseline, 3 months, 6 months. 9 months, 12 months, 15 months
  Items adapted from the National Survey of Veterans and prior studies examining health and social service use among individuals experiencing IPV, particularly in terms of VA and non-VHA psychosocial health services (e.g., mental health, housing, domestic violence agencies). The number and types of psychosocial treatment services will be examined.
VHA health care use | 12 months before baseline, 12 months after baseline
  VHA health care use will be extracted from the electronic medical records. The types and number of services used, particularly psychosocial health services, will be examined.
Treatment satisfaction | 3 months
  Treatment satisfaction will be assessed using the 8-item Client Satisfaction Questionnaire-8 (CSQ-8). Possible scores range from 8 to 32, with higher values indicating higher treatment satisfaction.
Perceived Benefits/Harms | 3 months
  Perceived benefits/harms from participating in the interventions will be measured using 6 items adapted from prior studies. Possible responses on a Likert scale range from 1= strongly disagree to 5 = strongly agree, with item 4 reverse scored. Individual item scores and total scores will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Iverson, PhD, Principal Investigator — V Boston Healthcare System, BU CASchool Medicine Psychiatry; Melissa Dichter, PhD MSW, Principal Investigator — VA Philadelphia Healthcare System
Locations (3):
- United States (3):
  - VA Boston Healthcare System, Boston, Massachusetts
  - VA Minneapolis Healthcare System, Minneapolis, Minnesota
  - VA Philadelphia Healthcare System, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No